CLINICAL TRIAL: NCT00669240
Title: Champix Observational Investigation In The Cessation of Smoking
Brief Title: Varenicline Observational Investigation In The Cessation of Smoking
Acronym: CHOICES
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051085
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1. Non-interventional: Patients prescribed varenicline in a non interventional manner.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — According to the approved Summary of Product Characteristics (SmPC), patients will be required to orally take 0.5 mg once daily for the first 3 days and titrate up to 0.5 mg twice daily for days 4 - 7. From day 8 to the end of treatment patients should take 1 mg twice daily. Patients who cannot tolerate adverse effects of Champix may have the dose lowered temporarily or permanently to 0.5 mg twice daily. Patients should be treated for 12 weeks. Treatment should start 1 - 2 weeks prior to quitting smoking.
  Other Names: Champix, Chantix, CP-526,555

SUMMARY:
The purpose of this study is to determine the safety and efficacy of varenicline in the real-world environment of smokers attending primary care in routine clinical practice with the addition of being offered behavioral support "Life REWARDS"TM. This is a non-interventional study.

DETAILED DESCRIPTION:
Sampling Method Details: Patients as they come to surgeries for smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients enrolled should be of legal adult age who regularly smoke and of which the main tobacco product is cigarettes.
* The patients must be willing to make an attempt to stop smoking.

Exclusion Criteria:

* All patients enrolled should meet the usual prescribing criteria for varenicline as per SmPC and should be entered into the trial at the Investigators discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled should be of legal adult age who regularly smoke and of which the main tobacco product is cigarettes. The patients must be willing to make an attempt to stop smoking.
  All patients enrolled should meet the usual prescribing criteria for varenicline as per SmPC and should be entered into the trial at the Investigators discretion.
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- Belgium (24):
  - Pfizer Investigational Site, Alleur
  - Pfizer Investigational Site, Beerse
  - Pfizer Investigational Site, Braine-le-Comte
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Deinze
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Habay-la-Neuve
  - Pfizer Investigational Site, Halen
  - Pfizer Investigational Site, Jette
  - Pfizer Investigational Site, Kortessem
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Libramont-Chevigny
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Moerkerke
  - Pfizer Investigational Site, Monceau-sur-Sambre
  - Pfizer Investigational Site, Moorsel
  - Pfizer Investigational Site, Namur
  - Pfizer Investigational Site, Rijkevorsel
  - Pfizer Investigational Site, Vedrin
  - Pfizer Investigational Site, Vilvoorde
  - Pfizer Investigational Site, Yvoir
  - Pfizer Investigational Site, Zedelgem
- Greece (10):
  - Pfizer Investigational Site, Cholargós, Athens
  - Pfizer Investigational Site, Ilisia, Athens
  - Pfizer Investigational Site, Marousi, Athens
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Eksochi, Thessaloniki
  - Pfizer Investigational Site, Alexandroupoli
  - Pfizer Investigational Site, Ioannina
  - Pfizer Investigational Site, Kavala
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Thessaloniki
- Hungary (9):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Eger
  - Pfizer Investigational Site, Érd
  - Pfizer Investigational Site, Farkasgyepű
  - Pfizer Investigational Site, Hatvan
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Siófok
  - Pfizer Investigational Site, Szombathely
  - Pfizer Investigational Site, Zalaegerszeg
- Slovenia (6):
  - Pfizer Investigational Site, Cerknica
  - Pfizer Investigational Site, Domžale
  - Pfizer Investigational Site, Jesenice
  - Pfizer Investigational Site, Kranj
  - Pfizer Investigational Site, Ljubljana
  - Pfizer Investigational Site, Maribor

REFERENCES:
- [Derived] Boudrez H, Hoengenaert JP, Nackaerts K, Messig M, Metcalfe M. Predictors of quit success in Belgian participants of a varenicline observational smoking cessation study. Acta Clin Belg. 2013 Jan-Feb;68(1):37-42. doi: 10.2143/ACB.68.1.2062718. PMID 23627193
- [Derived] Gratziou C, Gourgoulianis K, Pataka PA, Sykara GD, Messig M, Raju S. Varenicline as a smoking cessation aid in a Greek population: a subanalysis of an observational study. Tob Induc Dis. 2012 Feb 2;10(1):1. doi: 10.1186/1617-9625-10-1. PMID 22300423
- [Derived] Boudrez H, Gratziou C, Messig M, Metcalfe M. Effectiveness of varenicline as an aid to smoking cessation: results of an inter-European observational study. Curr Med Res Opin. 2011 Apr;27(4):769-75. doi: 10.1185/03007995.2011.557718. Epub 2011 Feb 4. PMID 21294601

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: According to the approved Summary of Product Characteristics (SmPC), participants were required to take 0.5 milligram (mg) orally once daily for the first 3 days and titrate up to 0.5 mg twice daily for days 4-7. From Day 8 to the end of treatment, participants should have taken 1 mg twice daily. Participants who cannot tolerate adverse effects of Champix could have the dose lowered temporarily or permanently to 0.5 mg twice daily. Participants were to be treated for 12 weeks, at which time a maintenance period of 12 weeks could be prescribed. Treatment was to start 1-2 weeks prior to quitting smoking.
Period: Overall Study
Arm/Group | Varenicline
Started | 567
Assigned to Treatment | 566
Received Treatment | 551
Completed | 402
Not Completed | 165
Not completed — Lack of Efficacy | 33
Not completed — Withdrawal by Subject | 42
Not completed — Lost to Follow-up | 34
Not completed — Adverse Event | 21
Not completed — Other | 19
Not completed — Enrolled but not treated | 15
Not completed — Enrolled but no dosing record | 1

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 551
Age, Customized [Number; unit: participants]
  <55 years | 415
  >=55 years and <=65 years | 107
  >65 years | 26
  Unspecified | 3
Sex/Gender, Customized [Number; unit: participants]
  Male | 295
  Female | 248
  Unspecified | 8
Number of years participants smoked [Mean (Full Range); unit: years] | 27.0 [2.0 to 60.0]
Average number of cigarettes participants smoked per day [Mean (Full Range); unit: cigarettes per day] | 25.3 [5.0 to 100.0]
Number of participants with quit smoking history [Number; unit: participants] — Number of participants who provided at least one reason for prior relapse (= number of participants with at least one prior quit smoking attempt)
  participants | 426
Total score on the Fagerstrom Test for Nicotine Dependence [Mean (Full Range); unit: scores on a scale] — The self-administered Fagerstrom Test for Nicotine Dependence questionnaire assesses level of nicotine dependence. Total score: 0-2=very low dependence; 3-4=low dependence; 5=medium dependence; 6-7=high dependence; 8-10=very high dependence.
  scores on a scale | 6.1 [0.0 to 10.0]
Reasons for quitting smoking [Number; unit: participants] — Each participant was asked to supply the top 2 reasons for giving up smoking this time; not all participants supplied 2 reasons.
  participants
    Family / friends | 255
    Health reasons | 495
    Money / cost | 159
    Body image / appearance | 84
    Smoking ban in public places | 35
Smoking-related concurrent illnesses and cardiovascular risk factors [Number; unit: participants] — Some participants may have had more than 1 condition and may be represented in more than 1 category, and some participants may not have had any condition.
  participants
    Diabetes | 31
    Raised cholesterol | 114
    Hypertension | 110
    Cardiovascular disease | 54
    Chronic obstructive pulmonary disease (COPD) | 100
    Lung cancer | 10
    Epilepsy | 9
    Psychiatric disorders (excluding depression) | 18
    Depression | 52
Source of reimbursement [Number; unit: participants] — Source of funding for the cost of varenicline treatment. Some participants listed more than one source of funding and are represented in more than 1 category.
  participants
    Public insurance | 214
    Private insurance | 2
    Self-payment | 353

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: Non-serious AEs are any untoward medical occurrence in a clinical investigation (subject administered a product or medical device) observed or volunteered through 7 days after the last dose of study drug regardless of suspected causal relationship; SAEs are any untoward medical occurrence that results in death; is life-threatening; requires hospitalization or prolongation of hospitalization; results in disability or incapacity; congenital anomaly or birth defect observed or volunteered through 28 days after the last dose of study drug, regardless of suspected causal relationship.
Time Frame: Baseline through Week 12 or Week 24
Population: Safety population, which is identical to the all-subjects population: all enrolled subjects who received at least 1 dose (including partial doses) of varenicline; Week 24 if a maintenance period was prescribed.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  Non-serious AEs | 131
  SAEs | 7

2. Secondary Outcome: Number of Participants Whose Smoking Status Was Known at the End of 12 Weeks
Description: Number of participants who were determined to be a responder or a non-responder at the specified time point. (Responders are participants who answered "no" to both of the following 2 questions, and non-responders are participants who answered "yes" to at least 1 of the following 2 questions, on the Nicotine Use Inventory (NUI): 1) Has the subject smoked any cigarettes (even a puff) in the last 7 days? 2) Has the subject used any other tobacco products (for example, pipe, cigars, snuff, chew) in the last 7 days?)
Time Frame: Week 12
Population: All-subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  Responders | 356
  Non-responders | 135

3. Secondary Outcome: Number of Participants in Belgium Whose Smoking Status Was Known at the End of 12 Weeks and 24 Weeks
Description: Number of participants in Belgium who were determined to be a responder or a non-responder at the specified time point. (Responders are participants who answered "no" to both of the following 2 questions, and non-responders are participants who answered "yes" to at least 1 of the following 2 questions, on the Nicotine Use Inventory (NUI): 1) Has the subject smoked any cigarettes (even a puff) in the last 7 days? 2) Has the subject used any other tobacco products (for example, pipe, cigars, snuff, chew) in the last 7 days?)
Time Frame: Week 12 and Week 24
Population: All-subjects population in Belgium
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 226
participants
  Week 12 Responders | 138
  Week 12 Non-responders | 41
  Week 24 Responders | 103
  Week 24 Non-responders | 34

4. Secondary Outcome: Number of Treatment Responders at Week 12
Description: Responders are participants who answered "no" to both of the following 2 questions on the Nicotine Use Inventory (NUI): 1) Has the subject smoked any cigarettes (even a puff) in the last 7 days? 2) Has the subject used any other tobacco products (for example, pipe, cigars, snuff, chew) in the last 7 days?
Time Frame: Week 12
Population: All-subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants | 356

5. Secondary Outcome: Number of Treatment Responders in Belgium at Week 12 and at Week 24
Description: as for outcome 4
Time Frame: Week 12 and Week 24
Population: All-subjects population in Belgium
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 226
participants
  Week 12 | 138
  Week 24 | 103

6. Secondary Outcome: Number of Participants With Smoking Cessation Assessments at Weekly Intervals From Week 3 Through Week 11
Description: Assessment of smoking cessation (ie, not a single puff) in previous 7 days, at time points of routine review of patients per local clinical practice.
Time Frame: Weeks 3, 4, 5, 6, 7, 8, 9, 10, and 11
Population: All-subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  Week 3 | 105
  Week 4 | 129
  Week 5 | 84
  Week 6 | 65
  Week 7 | 50
  Week 8 | 45
  Week 9 | 38
  Week 10 | 18
  Week 11 | 23

7. Secondary Outcome: Number of Treatment Responders at Weekly Intervals From Week 3 Through Week 11
Description: Responders are participants who answered "no" to the following 2 questions: 1) Has the subject smoked any cigarettes (even a puff) in the last 7 days? 2) Has the subject used any other tobacco products (for example, pipe, cigars, snuff, chew) in the last 7 days? Assessment conducted at specified time points only when usual for the local clinical practice.
Time Frame: Weeks 3, 4, 5, 6, 7, 8, 9, 10, and 11
Population: All-subjects population; n=number of participants in the All-subjects population with analyzable data (responders and non-responders) who were assessed for smoking cessation at the time point (per local clinical practice) .
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  Week 3 (n=105) | 65
  Week 4 (n=129) | 89
  Week 5 (n=84) | 62
  Week 6 (n=65) | 50
  Week 7 (n=50) | 43
  Week 8 (n=45) | 35
  Week 9 (n=38) | 28
  Week 10 (n=18) | 11
  Week 11 (n=23) | 19

8. Secondary Outcome: Number of Participants for Whom a Maintenance Period of Varenicline Was Prescribed at the End of Week 12
Description: A maintenance period was an additional period of varenicline treatment that could be prescribed at Week 12 by the attending primary care physician in routine clinical practice
Time Frame: Week 12
Population: All-subjects population
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants | 60

9. Secondary Outcome: Number of Participants Who Received Varenicline, by Duration of Treatment in Days
Time Frame: Baseline through Week 12 or Week 24
Population: All-subjects population; Week 24 if a maintenance period was prescribed.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  <=1 day | 3
  2-7 days | 8
  8-14 days | 19
  15-28 days | 48
  29-60 days | 85
  61-90 days | 280
  >=91 days | 108

10. Secondary Outcome: Number of Participants Who Registered With LifeREWARDS On-line Behavioral Support Program
Description: Number of participants who answered 'yes' to the question "Did you register with LifeREWARDS?" (LifeREWARDS not available in Greece.)
Time Frame: Week 12
Population: All-subjects population; n=number of participants with analyzable data at observation (responded to the question at the last study visit).
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 551
participants
  Belgium (n=194) | 65
  Greece (n=98) | 0
  Hungary (n=107) | 3
  Slovenia (n=15) | 2

11. Secondary Outcome: Minnesota Nicotine Withdrawal Scale (MNWS) Subscale Scores for Participants in Belgium
Description: Self-administered rating of intensity of nicotine withdrawal symptoms over past 24 hours; consists of 9 questions (urge to smoke, depressed mood, irritability, anxiety, difficulty concentrating, restlessness, increased appetite, difficulty going to sleep, difficulty staying asleep), each rated 0-4 (0=not at all, 1=slight, 2=moderate, 3=quite a bit, 4=extreme). Subscales: Negative affect domain (average of items 2-5); Insomnia domain (average of items 8 and 9); Urge to smoke (item 1); Restlessness (item 6); Increased appetite (item 7). Range 0-4 (higher score=greater intensity of symptoms)
Time Frame: Week 7 and Week 13 or 14 (Week 13/14)
Population: All subjects population in Belgium; n=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline
Number analyzed (Participants) | 226
scores on a scale
  Week 7: Negative affect domain (n=137) | 0.7 (0.7)
  Week 13/14: Negative affect domain (n=137) | 0.6 (0.7)
  Week 7: Insomnia domain (n=137) | 0.8 (1.0)
  Week 13/14: Insomnia domain (n=137) | 0.5 (0.8)
  Week 7: Urge to smoke (n=137) | 1.1 (1.0)
  Week 13/14: Urge to smoke (n=137) | 0.8 (0.9)
  Week 7: Restlessness (n=137) | 0.8 (1.0)
  Week 13/14: Restlessness (n=137) | 0.6 (0.9)
  Week 7: Increased appetite (n=134) | 1.1 (1.2)
  Week 13/14: Increased appetite (n=134) | 0.9 (1.1)

ADVERSE EVENTS:
Time Frame: 12 weeks and up to 24 weeks for participants presribed maintenance period
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 7/551
Other Adverse Events (participants affected / at risk) | 93/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=551)
Cardiovascular disorder (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mental disorder (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=551)
Abdominal pain upper (Gastrointestinal disorders) | 9
Gastritis (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 49
Fatigue (General disorders) | 7
Abnormal dreams (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 16
Sleep disorder (Psychiatric disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.